CLINICAL TRIAL: NCT04465305
Title: A Randomized Controlled Study of Nerve Root Sleeve Reinforcement and Reconstruction and Sacral Canopy for the Treatment of Sacral Canal Cysts
Brief Title: A Randomized Controlled Study on the Treatment of Sacral Canal Cysts With Sacral Canal Reinforcement
Acronym: ARCSTSCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUTHNSD
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2020-07

CONDITIONS: Tarlov Cysts
Keywords: tarlov cysts surgery
MeSH Terms: conditions — Tarlov Cysts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enraped group (Experimental): patients with a new treatment of tarlov cysts
  Interventions: Procedure: entraped treatment; Procedure: plasty treatment
- plasty group (Active Comparator): patients with traditional treatment of tarlov cysts
  Interventions: Procedure: plasty treatment

INTERVENTIONS:
Procedure: entraped treatment — patients with tarlov cysts treated by entraped and plasty nerve root
  Other Names: plasty treatment
  Arms: enraped group
Procedure: plasty treatment — patients with tarlov cysts treated by plasty nerve root

SUMMARY:
The subject will treat 68 patients with symptomatic sacral canal cysts as the research object, and adopt a randomized controlled research method, respectively, using two methods of reinforcement and reconstruction of the nerve root sleeve, sacroplasty and nerve root sleeve plasty, and observed the operation of the patient Complications, preoperative and postoperative short-term and long-term VAS pain scores, JOA neural function scores, and changes in cyst size on imaging examinations, to evaluate the safety of nerve root sleeve reconstruction and sacroplasty in reducing the safety of postoperative cyst recurrence Sex and effectiveness, so as to further improve the surgical treatment of sacral canal cysts, improve the curative effect, and formulate the operation specifications for the treatment of sacral canal cyst

DETAILED DESCRIPTION:
In this subject, a cohort observation method was used to observe 52 patients with two types of surgical removal of hematoma in the basal ganglia under the guidance of frontal ultrasound through keyhole neuroendoscopy and microsurgery for hematoma removal under the guidance of frontal ultrasound. They were divided into endoscopic surgery group and microsurgery. In the endoscopic surgery group, 26 cases were treated with keyhole neuroendoscopy under the guidance of frontal ultrasound for hematoma removal in the basal ganglia area, and 26 cases in the microsurgery group were treated by craniotomy microsurgery hematoma removal surgery. Observe the removal rate of surgical hematoma in the two groups And the safety of the operation and the GCS score, GOS score and MRI examination of nerve fiber damage and postoperative complications at 1 week, 1 month, and 3 months after the operation. Observe and analyze the improvement of the hematoma clearance rate in the endoscopic surgery group. And whether it has an advantage in terms of efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic nerve root cysts diagnosed by MRI
2. Intact cyst capsule, no defect of sacral canal lamina
3. No other diseases of nervous system, pelvic floor and important organs
4. Agree inclusion

Exclusion Criteria:

a ) Non-radiculent cysts or asymptomatic cysts b) Cysts cause severe bone erosion to lamina resorption c) Combined with other diseases of nervous system, pelvic floor and important organs d) Disagree to join e) Cannot complete follow-up -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
recurrent rate of tarlov cysts | 1 year
  patents who recurrent postoperation

CONTACTS AND LOCATIONS:
Overall Officials: liu bin, Study Chair — Peking University Third Hospital; wang zhenyu, Study Director — Peking University Third Hospital; xie jinchen, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No